CLINICAL TRIAL: NCT04260958
Title: Remote Exercise SWEDEHEART Study - a Multicentre Registry-based Cluster Randomized Crossover Clinical Trial (RRCT)
Brief Title: Remote Exercise SWEDEHEART Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Maria Bäck, Associate professor, physiotherapist, Sahlgrenska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U-2018-312
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Infarction
Keywords: Exercise-based cardiac rehabilitation; Secondary prevention; EHealth; Telerehabilitation; Physical fitness; Health-related quality of life; cost-effectiveness
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: CR centers will be cluster randomized and start as either the intervention or control center. Patients at intervention centers will be offered remote video exCR (first-hand option), usual care centre-based exCR or a combination of these two exercise modes. At control centers, patients will be offered usual care centre-based exCR only. The duration of each time period for each center will be 15 months and then cross-over will occur, so that intervention centers become control centers and the other way around. At intervention centers, patients participating in remote exCR will finish their 3-month exercise period, but no new patients will be offered remote exCR after the cross-over has occurred.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention center (Experimental): Patients at intervention centers will be offered remote video exCR (first-hand option), usual care centre-based exCR or a combination. The exercise program (remote/centre-based) will be standardized and performed for totally 60 minutes, 2 times a week for 3 months. Exercise will be individually prescribed and progressed by physiotherapists in accordance with guidelines. Patients will also be asked to perform one additional session of at least 30 min aerobic exercise per week, at intensity level 13-15 according to Borg RPE-scale.
  Interventions: Other: Exercise-based cardiac rehabilitation
- Control (No Intervention): At control centers, patients will be offered usual care centre-based exCR only. Patients will also be asked to perform one additional session of at least 30 min aerobic exercise per week, at intensity level 13-15 according to Borg RPE-scale.

INTERVENTIONS:
Other: Exercise-based cardiac rehabilitation — The exercise program (remote/centre-based) will be standardized. An exCR-program is defined as at least 24 supervised sessions, with a total session length of 60 minutes, for at least 3 months, with possibility to complete missed sessions the 4th month. Each exercise session includes at least 20 min of aerobic exercise, intensity 13-17 on Borg´s rating of perceived exertion (RPE)-scale ≈ 60% - 85% of VO2max or 70 - 95% of maximal heart rate. In addition, each exercise session includes 1-3 sets of 8-10 upper and/or lower limb exercises in 10-15 repetitions, 40-80% of 1 repetition maximum. Attending ≥75% of the 24 sessions over a 4-month period will be considered as successful.
  Arms: Intervention center

SUMMARY:
The overall aim of the study is to evaluate if remote video exercise-based cardiac rehabilitation (exCR), offered as an alternative to centre-based exCR, can increase participation in exCR sessions post myocardial infarction (MI).

DETAILED DESCRIPTION:
Due to the covid-19 pandemic, this study will be performed in two steps:

1). National feasibility and safety study. 2). National multicenter registry-based cluster randomized crossover clinical trial (RRCT).

1. In the feasibility study, patients will be offered remote exCR at all participating sites until the peak of the pandemic has been achieved and care goes back to normal. The feasibility study will include patients until Aug 2022.
2. CR centers (not patients) will be cluster randomized to either the intervention or control. Patients at intervention centers will be offered remote exCR, usual care centre-based exCR, or a combination of both modes, as self-preferred choice. At control centers, patients will be offered usual care centre-based exCR only. The duration of each time period for each center will be 15 months. Long-term follow-up will be performed 1 year and 3 years after the index cardiac event.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of type 1 myocardial infarction (AMI)
* Age 18-79 years at discharge from hospital

Exclusion Criteria:

* Patients with incomplete coronary revascularization defined as at least one remaining hemodynamically significant stenosis
* Severe valve or structural heart disease
* Severe heart failure (NYHA III - IV)
* Serious arrythmias
* Inability to understand Swedish
* No internet access at home (only applicable for patients in the intervention group who wants to perform remote exCR)
* Pathological exercise test indicating high risk for adverse events during exCR
* More than 6 months between discharge form hospital and screening
* Any other condition that may interfere with the possibility for the patient to comply with the study protocol

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean number of exCR sessions | 3-4 months
  The primary outcome is the mean number of EBCR sessions (center based or remote) during 0-4 months (from start of the EBCR program) for patients at a center during each randomization period. Eligible patients that have not started the EBCR program within 6 months of screening will be counted as 0 sessions. Attending ≥75% of the 24 recommended sessions over a 4-month period will be considered as completion, and proportion completers will be presented in a supportive responder analysis.

SECONDARY OUTCOMES:
Submaximal exercise capacity | 3-4 months
  Bicycle ergometer test according to the WHO-protocol with an increased workload of 25W every 4.5 minutes. The exercise test is discontinued at Borg RPE 17 and/or dyspnea 7 at Borg´s CR-10 scale.
Muscular endurance tests | 3-4 months
  Unilateral isotonic shoulder flexion (maximum number of repetitions) and a unilateral isotonic heel lift (maximum number of repetitions)
Self-reported physical activity and exercise | 3-4 months
  Two questions on physical activity and exercise during the latest week according to Haskell´s questionnaire (Min:0, Max:7). Ordinal scale, number of days.
Self-reported physical activity and exercise Haskell | 3-4 months
  Haskell´s questionnaire (Min:0, Max:7). A high score means higher level of physical activity and exercise.
Self-reported physical capacity | 3-4 months
  Visual analog scale, (100=best possible physical capacity, 0=worst possible physical capacity), a dichotomous question: Do you experience any limitation in everyday life due to your current physical capacity? (yes vs no). If yes: multiple choice on reasons
Health-related quality of life EQ5D | 3-4 months
  Euro Quality of Life (EQ-5D 3L). The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. A high score indicates better Health.
Health-related quality of life VAS | 3-4 months
  Euro Quality of Life VAS. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state'(100) and 'Worst imaginable health state' (0)
Kinesiophobia (fear of movement) | 3-4 months
  Tampa Scale for Kinesiophobia Heart (17 items, ordinal scale 1-4) 1, strongly disagree, 4, strongly agree. A higher score is means higher values of kinesiophobia (worse).
Self-efficacy for Exercise Scale | 3-4 months
  Self-efficacy for Exercise Scale. 9 items, ordinal scale. 0=not Confident, 10=very Confident. Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise
Self-reported perceptions on exercise | 3-4 months
  Patient´s perceptions of remote exCR or centre-based exCR. 1, strongly disagree, 4, strongly agree. This questionnarie is designed by the authors. High score, better outcome.
Cost-effectiveness | End of study
  A cost-effectiveness analysis will be performed in order to estimate the cost per quality-adjusted life-year (QALY) associated with the intervention compared with control. Healthcare costs associated with investigated treatments will be assessed by extracting resource use from the relevant registries, and QALYs will be determined by combining survival status and the quality-of-life measurements provided by the EQ-5D-3L instrument.
Socio-economic evaluation | 6 years
  Data from Statistics Sweden will be used to evaluate study results in relation to socio-economic data
Number of Cardiovascular events | 1 and 3 years after the last patient visit
  All-cause mortality, cardiovascular mortality, recurrent hospitalization for ACS, heart failure hospitalization, stroke and repeat coronary revascularization, reported in SWEDEHEART, the National Patient Registry and the Cause of Death Register will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Back, Ass Prof, Principal Investigator — Sahlgrenska University Hospital; Stefan James, Prof, Study Chair — Uppsala Clinial Research Center
Locations (26):
- Sweden (26):
  - Södra Älvsborg Hospital, Borås
  - Mälarsjukhuset, Eskilstuna
  - Falun hospital, Falun
  - Gällivare Hospital, Gällivare
  - Gävle Hospital, Gävle
  - Angered Hospital, Gothenburg
  - Sahlgrenska University Hospital Östra, Gothenburg
  - Sahlgrenska University Hospital, Gothenburg
  - Hässleholm Hospital, Hässleholm
  - Jönköping Ryhov hospital, Jönköping
  - Kalix hospital, Kalix
  - Kalmar Hospital, Kalmar
  - Kungälv Hospital, Kungälv
  - Lindesberg Hospital, Lindesberg
  - Linköping University Hospital, Linköping
  - Ljungby Hospital, Ljungby
  - Sunderbyn hospital, Luleå
  - Skåne University hospital, Lund
  - Skåne University Hospital Malmö, Malmo
  - Östersund hospital, Östersund
  - Södertälje Hospital, Södertälje
  - Capio St Göran Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Sundsvall hospital, Sundsvall
  - Uppsala University Hopsital, Uppsala
  - Värnamo hospital, Värnamo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Back M, Leosdottir M, Ekstrom M, Hambraeus K, Ravn-Fischer A, Oberg B, Ostlund O, James S. The remote exercise SWEDEHEART study-Rationale and design of a multicenter registry-based cluster randomized crossover clinical trial (RRCT). Am Heart J. 2023 Aug;262:110-118. doi: 10.1016/j.ahj.2023.04.014. Epub 2023 Apr 25. PMID 37105430
- [Derived] Back M, Leosdottir M, Ekstrom M, Hambraeus K, Ravn-Fischer A, Borg S, Brosved M, Flink M, Hedin K, Lans C, Olovsson J, Urell C, Oberg B, James S. Feasibility, safety and patient perceptions of exercise-based cardiac telerehabilitation in a multicentre real-world setting after myocardial infarction-the remote exercise SWEDEHEART study. Eur Heart J Digit Health. 2025 Mar 4;6(3):508-518. doi: 10.1093/ehjdh/ztaf014. eCollection 2025 May. PMID 40395424